CLINICAL TRIAL: NCT04632953
Title: Long-Chain Fatty Acid Oxidation Disorders In-Clinic Disease Monitoring Program (LC-FAOD DMP)
Brief Title: Long-Chain Fatty Acid Oxidation Disorders In-Clinic Disease Monitoring Program
Status: Active, not recruiting | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX007-CL401
Record Dates: First submitted 2020-11-09; First posted 2020-11-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Long-chain Fatty Acid Oxidation Disorders (LC-FAOD)
Keywords: CACT Deficiency; Carnitine Acylcarnitine Translocase Deficiency; CPT1; CPT2; Carnitine Palmitoyltransferase Deficiencies; VLCAD; Very Long Chain Acyl Coa Dehydrogenase Deficiency; LCHAD Deficiency; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; TFP Deficiency; Trifunctional Protein Deficiency
MeSH Terms: conditions — Carnitine-Acylcarnitine Translocase Deficiency; VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Previously Treated with Triheptanoin: Patients who have been previously treated with triheptanoin in clinical studies: UX007-CL201 (NCT01886378), UX007-CL202 (NCT02214160), UX007-CL302 (2022-001539-10), Investigator Sponsored Trials (ISTs), or UX007-EAP (NCT03773770).
  Interventions: Other: No Intervention
- Cohort 2: Currently or Previously Treated with Triheptanoin: New patients enrolling into the DMP currently or previously treated with triheptanoin (excluding those in Cohort 1).
  Interventions: Other: No Intervention
- Cohort 3: Triheptanoin Naïve: New patients enrolling into the DMP with no exposure to triheptanoin (naïve).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The primary objective of this study is to assess the long-term safety, including pregnancy, infant, and lactation outcomes, of patients with LC-FAOD who are enrolled in the DMP.

DETAILED DESCRIPTION:
The LC-FAOD Disease Monitoring Program (DMP) is an international, long-term, retrospective and prospective outcomes study aiming to collect safety and effectiveness data for triheptanoin and the natural history of LC-FAOD for a study duration of up to 10 years from adult and pediatric patients with LC-FAOD, with any previous disease management, regardless of prior treatment with triheptanoin, those who have previously participated in triheptanoin clinical trials, and those who received triheptanoin through an Expanded Access Program (EAP).

Patients enrolling in the LC-FAOD DMP will be managed at the discretion of their physicians and may or may not be treated with triheptanoin during the course of the study. Patients will have access to triheptanoin only through authorized commercial use (if approved in their country) or available EAP but not from the LC-FAOD DMP itself.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of any LC-FAOD subtype. Diagnosis must be confirmed by results of acylcarnitine profiles and/or genetic testing results obtained from medical records or equivalent documentation.
* Willing and able to comply with all study procedures.
* Willing and able to provide consent or, if a minor, provide assent and informed consent by their legally authorized representative.
* Females of childbearing potential who become pregnant during the study will be invited to remain in the study. Pregnant females with LC-FAOD will be informed of the study and invited to enroll.

Exclusion Criteria:

* Presence of a concurrent disease or condition that would interfere with study participation or affect patient's safety in the opinion of the Investigator.
* Presence or history of any condition that, in the view of the Investigator, places the patient at high risk of not completing the study or would affect the interpretation of study results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 150 patients, either treated or untreated with triheptanoin, will be enrolled for this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Long-Term Safety of Patients With LC-FAOD as Assessed by Incidence, Severity, and Frequency of Serious Adverse Events (SAEs) and Adverse Events (AEs) in Pregnant and Lactating Patients with LC-FAOD | 10 Years
Long-Term Safety of Patients With LC-FAOD as Assessed by Outcomes of Pregnancy in Patients with LC-FAOD | 10 Years
Long-Term Safety of Patients With LC-FAOD as Assessed by Incidence, Frequency, and Severity of SAEs and AEs During the First Year of Life in Infants Born to Study Participants | 10 Years
Long-Term Safety of Patients With LC-FAOD as Assessed by Incidence of SAEs Assessed as Related to Triheptanoin Treatment by Study Investigator | 10 Years
Long-Term Safety of Patients With LC-FAOD as Assessed by Incidence of All Colon Cancer or Gastrointestinal (GI) Cancer, GI Dysplasia, and GI Neoplasia, SAEs and AEs Reported for All Patients With LC-FAOD | 10 Years

SECONDARY OUTCOMES:
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Major Clinical Events (MCEs) | 10 Years
  Frequency and duration of MCEs including events of rhabdomyolysis, cardiomyopathy, hypoglycemia, and other disease complications
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by At-Home Clinical Events (HCEs) | 10 Years
  Frequency and duration of HCEs including events of hypoglycemia, rhabdomyolysis, cardiomyopathy, and other disease complications
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Mortality | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Height | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Weight | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Head Circumference | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Body Mass Index (BMI) | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Distance Travelled in the 12-Minute Walk Test (12MWT) | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Change from Baseline in Echocardiogram (ECHO) Parameters: Left Ventricular Mass Index | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Change from Baseline in Echocardiogram (ECHO) Parameters: Left Ventricular Ejection Fraction | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Incidence and Type of Cardiac Arrhythmia | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Change from Baseline in Alanine Aminotransferase (ALT) | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Change from Baseline in Total Creatine Kinase (CK) | 10 Years
Long-Term Effectiveness of Triheptanoin in Patients With LC-FAOD as Assessed by Change from Baseline in Select Acylcarnitines | 10 Years
Dose-Response Relationship of Triheptanoin and Even-Chain MCT as Assessed by Incidence of MCEs and HCEs With Consideration of Diet | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by the Clinical Global Impression of Severity (CGI-S) Assessment | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by the Infant and Toddler Quality of Life (ITQOL) | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by the Medical Outcomes Study 10-Item Short Form (SF-10) | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by the Medical Outcomes Study 12-Item Short Form (SF-12 v2) | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by Medical Resource Utilization | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by Assistive Device Use | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by the Work Productivity Questionnaire | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by the School Impact Questionnaire | 10 Years
Impact of Triheptanoin on Patient- and Clinician-Reported Measures of Disease Severity and Burden as Assessed by Long-Term Complications of LC-FAOD | 10 Years
  May include retinopathy and peripheral neuropathy or other sensory and motor complications

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (16):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - CHEO (Children's Hospital Eastern Ontario), Ottawa, Ontario
  - SickKids (The Hospital for Sick Children), Toronto, Ontario

REFERENCES:
- See also: Ultragenyx Patient Advocacy/LC-FAOD Disease Information — https://ultrarareadvocacy.com/conditions-we-study/long-chain-fatty-acid-oxidation-disorders-lc-faod/
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/